CLINICAL TRIAL: NCT04422327
Title: An Open Label Study to Assess the Impact of 'COMBO' on Mood, Stress and Bowel Symptoms in Adults With Irritable Bowel Syndrome (IBS)
Brief Title: The Impact of a Combination of Bifidobacterium Longum 35624® and 1714™ Strains in Adults With Irritable Bowel Syndrome
Acronym: IBS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PrecisionBiotics Group Ltd. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFCRO-079
Record Dates: First submitted 2020-05-25; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: IBS - Irritable Bowel Syndrome; Depression, Anxiety
Keywords: Combination of probiotics; Bifidobacterium longum 35624®; Bifidobacterium longum 1714™; depression; anxiety; bowel symptoms; Irritable Bowel Syndrome (IBS); Sleep quality; Cognition; Safety
MeSH Terms: conditions — Irritable Bowel Syndrome; Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Open label study, with intervention period followed by follow-up (wash out) period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic capsule (Experimental): The participants consume one probiotic capsule a day for 8 weeks
  Interventions: Dietary Supplement: Probiotic capsule

INTERVENTIONS:
Dietary Supplement: Probiotic capsule — Each probiotic capsule contains 5 x 10^8 CFU B. longum 35624® and 5 x 10^8 CFU B. longum 1714™ with corn starch and magnesium stearate.
  The probiotic capsule will be supplied by PrecisionBiotics Ltd.

SUMMARY:
This study aimed to assess the impact of consumption of COMBO, a combination product of two Bifidobacterium longum strains, on stress, mood and bowel symptoms in adults with Irritable Bowel Syndrome (IBS).

DETAILED DESCRIPTION:
This is an open label study designed to assess the impact on stress, mood and bowel symptoms & safety of COMBO, a combination of Bifidobacterium longum 35624® and Bifidobacterium longum 1714™ strains, when consumed once daily for 8 weeks, in adults with Irritable Bowel Syndrome (IBS). Volunteers will be screened according to the selection criteria in order to identify up to 40 female subjects, with recurrent abdominal pain/discomfort and mild to moderate stress/mood status. The study will involve 6 visits over an 18 to 20-week period [Screening period (Visit 1: week-2), Intervention period (Visit 2: week 0, Visit 3: week 4, Visit 4: week 8), and Follow-up/ Washout period (Visit 5: week 12, Visit 6: week 16)]. Participants will fill in daily and weekly eDiary from 1st visit onwards. Questionnaires will be administered from visit 2 to visit 6. Research blood and saliva will also be collected at these time points. Stool sample will be collected at Visit 2, 4, 5, 6.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

1. Be able to give written informed consent,
2. Be a Caucasian female, between 18 and 55 years of age,
3. Subject has Irritable Bowel Syndrome according to the Rome III Diagnostic Criteria:

   Recurrent abdominal pain or discomfort** at least 3 days/month in the last 3 months associated with two or more of the following:

   i. Improvement with defecation

   ii. Onset associated with a change in frequency of stool

   iii. Onset associated with a change in form (appearance) of stool

   Criterion fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis

   ** "Discomfort" means an uncomfortable sensation not described as pain.
4. Subjects agree to complete symptom diaries and return completed diaries at all sessions,
5. Subjects with mild to moderate score (8-14) on the HADS-A and/or HADS-D questionnaire, Subjects will be excluded if there is greater than 1 point difference from the screening to baseline scores,
6. Be willing to refrain from taking any dietary supplements or other fermented foods that contain live bacteria during the study,
7. Be willing to refrain from taking any medications or preparations used in the therapy of IBS (herbal, dietary supplements, homeopathic preparations, etc.) during the study and from 4-weeks before the baseline visit,
8. Be willing to refrain from probiotic use 4 weeks before the baseline visit,
9. If using fiber supplements (e.g., Trifyba, Fybogel, Konsyl, Isogel, Regulan, Ispagel, Celevac, Normacol), the dose and regimen have remained stable for at least 30 days and the subject will continue the same dose and regimen throughout the length of the trial,
10. If using products that contain nicotine or caffeine, agrees to continue current usage levels throughout the length of the trial.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Are less than 18 and greater than 55 years of age at the time of consent,
2. Females are pregnant, lactating or wish to become pregnant during the study. Female subject is currently either of:

   * non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or any female who is surgically sterilized (via documented hysterectomy or bilateral tubal ligation). (For purposes of this study, postmenopausal is defined as one year without menses), OR
   * child bearing potential, the subject is eligible to enter and participate in this study if she is not lactating and has a negative urine pregnancy test at the screening visit, visit 2 and upon completion of the study at visit 7. The subject must also agree to one of the following methods of contraception:

     i. Complete abstinence from intercourse two weeks prior to administration of study drug, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study medication in cases where subject discontinues the study prematurely. (Subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit.) or,

   ii. has a male sexual partner who is surgically sterilized prior to the Screen Visit and is the only male sexual partner for that subject or,

   iii. sexual partner(s) is/are exclusively female or,

   iv. Oral contraceptives (either combined or progestogen only) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm. (Women of child-bearing potential using an oral contraceptive in combination with a double-barrier method of contraception are required to continue to use this form of contraception for 1 week following discontinuation of study medication).

   v. Use of double-barrier contraception, specifically, a spermicide plus a mechanical barrier (e.g. male condom, female diaphragm). The subject must be using this method for at least 1 week following the end of the study or,

   vi. Use of any intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1% per year. The subject must have the device inserted at least 2 weeks prior to the first Screen Visit, throughout the study, and 2 weeks following the end of the study,
3. Are hypersensitive to any of the components of the test product,
4. Consumption of Alflorex probiotic for 6 months,
5. Consumption of any type of yoghurts or probiotic-containing products in the 4 weeks prior to the baseline visit,
6. Subjects who have been on antibiotics during the past month,
7. Concurrent systemic disease and/or laboratory abnormalities considered by Investigators to be risky or that could interfere with data collection,
8. Subjects who have a significant acute or chronic coexisting illness [cardiovascular, history of co-existing gastrointestinal, and/or gynecological, and/or urologic pathology (eg., colon cancer, colitis, Crohn's, celiac, endometriosis, prostate cancer) or lactose intolerance,
9. Subjects with inflammatory disorders (e.g. chronic fatigue syndrome (CDC criteria), psoriasis, rheumatoid arthritis or any other inflammatory arthropathies),
10. Subjects who are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year),
11. Psychiatric diagnosis other than anxiety or depression,
12. Subjects who are on anti-depressants, anxiolytics, antipsychotics, anticonvulsants, centrally acting corticosteroids and/or opioid pain relievers in the last 6 months,
13. Subject has IBS symptoms that are predominantly related to menstruation,
14. Subject has a history of prior gastrointestinal surgery (apart from appendectomy),
15. Subjects who have had a previous cholecystectomy,
16. Subjects with a history of active cancer in the last 5 years (other than localized basal cell, squamous cell skin cancer or cancer in situ that has been resected),
17. Subjects with a history of drug and / or alcohol abuse at the time of enrolment,
18. Subject has a history of non-compliance,
19. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial,
20. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study,
21. Have a malignant disease or any concomitant end-stage organ disease.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Change in stress and mood, assessed by Hospital Anxiety and Depression Scale (HADS) scores | Assessed at baseline, 4 and 8 weeks of supplement intake, and 4 and 8 weeks post supplement intake.
  HADS gives HADS-A and HADS-D scores; minimum score for each is 0, maximum score is 21. Higher scores indicate worse stress/mood.

SECONDARY OUTCOMES:
Change in Subject Global Assessment (SGA) of IBS symptoms, assessed by weekly eDiary | Assessed weekly from baseline to 8 weeks post supplement intake.
  Participants answer the question: "Did you have adequate relief of your IBS symptoms over the past week?" Yes or No.
Change in Subject Global Assessment (SGA) of abdominal pain/discomfort, assessed by weekly eDiary | Assessed weekly from baseline to 8 weeks post supplement intake.
  Participants answer the question: "Did you have adequate relief of your abdominal pain and discomfort over the past week?" Yes or No.
Change in IBS-Symptom Severity Score (IBS-SSS) | Assessed at baseline, 4 and 8 weeks of supplement intake, and 4 and 8 weeks post supplement intake.
  IBS-SSS is a composite score of abdominal pain, number of days with abdominal pain, bloating/distension, satisfaction with bowel habits, and IBS-related quality of life (QoL). Scores range from 0 to 500, with higher scores indicating worse symptoms.
Change in stool frequency, assessed by daily eDiary | Assessed daily from baseline to 8 weeks post supplement intake.
  Daily diary of number of bowel movements.
Change in stool consistency (Bristol Stool Scale), assessed by daily eDiary | Assessed daily from baseline to 8 weeks post supplement intake.
  Daily diary of stool consistency of each bowel movement based on Bristol Stool Scale (Type 1-7).
Change in abdominal pain/discomfort, assessed by daily eDiary | Assessed daily from baseline to 8 weeks post supplement intake.
  Daily diary of Visual Analog Scale (VAS) of abdominal pain/discomfort.
Change in abdominal bloating/distension, assessed by daily eDiary | Assessed daily from baseline to 8 weeks post supplement intake.
  Daily diary of Visual Analog Scale (VAS) of abdominal bloating/distension.
Change in bowel movement urgency, assessed by daily eDiary | Assessed daily from baseline to 8 weeks post supplement intake.
  Daily diary of Visual Analog Scale (VAS) of bowel movement urgency.
Change in straining, assessed by daily eDiary | Assessed daily from baseline to 8 weeks post supplement intake.
  Daily diary of Visual Analog Scale (VAS) of straining.
Change in passage of gas, assessed by daily eDiary | Assessed daily from baseline to 8 weeks post supplement intake.
  Daily diary of Visual Analog Scale (VAS) of passage of gas.
Change in Visceral Sensitivity Index | Assessed at baseline, 4 and 8 weeks of supplement intake, and 4 and 8 weeks post supplement intake.
  Visceral Sensitivity Index (VSI) is a self-report measure of the gastrointestinal symptom-specific anxiety (GSA) of patients with IBS, in terms of cognitive, emotional and behavioral responses. Sum scores range from 0 to 75 with higher scores indicating more severe GI-specific anxiety.
Change in sleep quality, assessed by Pittsburgh Sleep Quality Index (PSQI) | Assessed at baseline, 4 and 8 weeks of supplement intake, and 4 and 8 weeks post supplement intake.
  PSQI global score: minimum score is 0, maximum score is 21. Higher scores indicate worse sleep quality.
Change in cognition, assessed by Visual Analogue Scales | Assessed at baseline, 4 and 8 weeks of supplement intake, and 4 and 8 weeks post supplement intake.
  This assessment measures individual question answers related to hedonic tone, anxiety and alertness.
Change in cognition, assessed by spatial span test | Assessed at baseline, 4 and 8 weeks of supplement intake, and 4 and 8 weeks post supplement intake.
  This test measures span length, errors, number of attempts and latency.
Change in cognition, assessed by Stockings of Cambridge test | Assessed at baseline, 4 and 8 weeks of supplement intake, and 4 and 8 weeks post supplement intake.
  This test measures problems solved in minimum moves, mean moves per n-move problem, initial thinking time per n-move problems and subsequent thinking time per n-move problems.
Change in cognition, assessed by Paired Associates Learning test | Assessed at baseline, 4 and 8 weeks of supplement intake, and 4 and 8 weeks post supplement intake.
  This test measures errors, trials, memory scores and stages completed.
Safety of the investigational product, assessed by number of participants with treatment-related adverse events | Assessed through study completion, an average of 6 months.
  Safety will be evaluated throughout the study on the basis of incidence of treatment-related serious and non-serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Murphy, PhD, Study Director — PrecisionBiotics Group Ltd.
Locations (1):
- Atlantia Food Clinical Trials Ltd., Cork, Ireland

IPD SHARING:
Plan to Share IPD: No